CLINICAL TRIAL: NCT02919163
Title: Systematically Assessing Effects of Colored Light on Humans With a Multi-modal Approach
Brief Title: Systematically Assessing Effects of Colored Light on Humans With a Multi-modal Approach (Substudy 6 of 7)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: COLOR10_f
Record Dates: First submitted 2016-08-24; First posted 2016-09-29 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Exposure to Man-made Visible Light
Keywords: cerebral oxygen metabolism; functional near-infrared spectroscopy; partial pressure of carbon dioxide; heart rate variability; blood pressure; affect; mood; respiration; systematic randomized cross-over study; systemic physiology; electro-dermal activity; pulse-respiratory quotient
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Visible light exposure Red 30 lux (Experimental): The participants will be exposed to incandescent light with a red color filter at a illuminance of 30 lux at eye level for 15 minutes. The colored light exposure will be preceded by sitting 8 minutes in darkness and followed by sitting 20 minutes in darkness.
  Interventions: Other: Visible light exposure
- Visible light exposure Red 120 lux (Experimental): The participants will be exposed to incandescent light with a red color filter at a illuminance of 120 lux at eye level for 15 minutes. The colored light exposure will be preceded by sitting 8 minutes in darkness and followed by sitting 20 minutes in darkness.
  Interventions: Other: Visible light exposure
- Visible light exposure Blue 30 lux (Experimental): The participants will be exposed to incandescent light with a blue color filter at a illuminance of 30 lux at eye level for 15 minutes. The colored light exposure will be preceded by sitting 8 minutes in darkness and followed by sitting 20 minutes in darkness.
  Interventions: Other: Visible light exposure
- Visible light exposure Blue 120 lux (Experimental): The participants will be exposed to incandescent light with a blue color filter at a illuminance of 120 lux at eye level for 15 minutes. The colored light exposure will be preceded by sitting 8 minutes in darkness and followed by sitting 20 minutes in darkness.
  Interventions: Other: Visible light exposure
- Visible light exposure Green 30 lux (Experimental): The participants will be exposed to incandescent light with a green color filter at a illuminance of 30 lux at eye level for 15 minutes. The colored light exposure will be preceded by sitting 8 minutes in darkness and followed by sitting 20 minutes in darkness.
  Interventions: Other: Visible light exposure
- Visible light exposure Green 120 lux (Experimental): The participants will be exposed to incandescent light with a green color filter at a illuminance of 120 lux at eye level for 15 minutes. The colored light exposure will be preceded by sitting 8 minutes in darkness and followed by sitting 20 minutes in darkness.
  Interventions: Other: Visible light exposure
- Visible light exposure White 30 lux (Experimental): The participants will be exposed to incandescent light with no color filter at a illuminance of 30 lux at eye level for 15 minutes. The colored light exposure will be preceded by sitting 8 minutes in darkness and followed by sitting 20 minutes in darkness.
  Interventions: Other: Visible light exposure
- Visible light exposure White 120 lux (Experimental): The participants will be exposed to incandescent light with no color filter at a illuminance of 120 lux at eye level for 15 minutes. The colored light exposure will be preceded by sitting 8 minutes in darkness and followed by sitting 20 minutes in darkness.
  Interventions: Other: Visible light exposure

INTERVENTIONS:
Other: Visible light exposure — Subjects will be exposed to visible colored light for 15 minutes. The visible light will be generated by incandescent white light bulbs and color filters.

SUMMARY:
NOTE: This is the sixth of in total 7 sub-studies related to the Ethics Committee of the Canton of Bern Ref. No. KEK-BE 2016-00674. This sub-study includes 50 participants and 8 arms, in total 350 participants will be assessed in all 7 sub-studies.

General study information: This is a randomized, cross-over, quantitative study, which investigates physiological variables, mood, and affect of healthy participants in response to colored light exposure. The Participants take part in 5-8 arms and are exposed to colored light only, or are additionally asked to solve cognitive tasks during the colored light exposure. Primary aim is to measure the change in several physiological variables, mood, and affect during colored light exposure of 15 or 45 minutes. The risk for the participants is negligible and comparable to the risk during daily life.

ELIGIBILITY:
Inclusion Criteria:

* Normal color vision
* Right handed
* Written informed consent

Exclusion Criteria:

* Smoking
* Any kind of diagnosed sleep disorder or neurological or psychiatric disorder in the last 3 months
* Acute severe traumas
* Chronic diseases with the necessity for medication
* Use of recreational drugs
* Regular intake of medication that would affect the outcome measures
* Regular excessive alcohol use (> 18 standard units / week)
* Transmeridian travel in the last month (crossed > 1 time zone border)
* Night shift word during the last month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2027-12-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2029-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral tissue oxygen saturation during colored light exposure compared with a baseline and a recovery period | 43 minutes (8 min baseline, 15 min colored light exposure, 20 min recovery)
Change in cerebral hemoglobin concentration during colored light exposure compared with a baseline and a recovery period | 43 minutes (8 min baseline, 15 min colored light exposure, 20 min recovery)
Change in variables of the heart rate variability during colored light exposure compared with a baseline and a recovery period | 43 minutes (8 min baseline, 15 min colored light exposure, 20 min recovery)
Change in variables of the electro-dermal activity during colored light exposure compared with a baseline and a recovery period | 43 minutes (8 min baseline, 15 min colored light exposure, 20 min recovery)
Change of the blood pressure during colored light exposure compared with a baseline and a recovery period | 43 minutes (8 min baseline, 15 min colored light exposure, 20 min recovery)
Change of the partial pressure of carbon dioxide during colored light exposure compared with a baseline and a recovery period | 43 minutes (8 min baseline, 15 min colored light exposure, 20 min recovery)
Change of the respiration rate during colored light exposure compared with a baseline and a recovery period | 43 minutes (8 min baseline, 15 min colored light exposure, 20 min recovery)
Change of the heart rate during colored light exposure compared with a baseline and a recovery period | 43 minutes (8 min baseline, 15 min colored light exposure, 20 min recovery)
Change of the pulse-respiratory quotient during colored light exposure compared with a baseline and a recovery period | 43 minutes (8 min baseline, 15 min colored light exposure, 20 min recovery)
  The pulse-respiratory quotient will be calculated as heart rate divided by the respiration rate.
Change of the arterial oxygen saturation during colored light exposure compared with a baseline and a recovery period | 43 minutes (8 min baseline, 15 min colored light exposure, 20 min recovery)

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Wolf, Prof. Dr., Principal Investigator — University of Bern
Locations (1):
- University of Bern, Institute of Complementary Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Access to research data and documents will be handled according to the Manifesto to advance Data Access and Research Transparency (DART) in Switzerland, formulated at the workshop on "Improving DART in Switzerland" in Bern, November 7th, 2014.

REFERENCES:
- [Background] Weinzirl J, Wolf M, Nelle M, Heusser P, Wolf U. Colored light and brain and muscle oxygenation. Adv Exp Med Biol. 2012;737:33-6. doi: 10.1007/978-1-4614-1566-4_5. No abstract available. PMID 22259078
- [Background] Weinzirl J, Wolf M, Heusser P, Nelle M, Wolf U. Effects of changes in colored light on brain and calf muscle blood concentration and oxygenation. ScientificWorldJournal. 2011 Jun 9;11:1216-25. doi: 10.1100/tsw.2011.118. PMID 21666991
- See also: Link to further information on the study — http://www.ikom.unibe.ch/forschung/fachbereiche/anthroposophisch_erweiterte_medizin/index_ger.html